CLINICAL TRIAL: NCT06918795
Title: Home-based, Digital Intervention to Increase Physical Activity in Patients With the Fontan Circulation
Brief Title: Fontan Fitness Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-022619; 1R61HL171110-01A1 (NIH)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Single-ventricle; Congenital Heart Disease
Keywords: Fontan; Single ventricle disease; exercise intervention; digital health; adolescents; randomized control trial
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Exercise Intervention (Experimental): The exercise intervention arm includes access to a digital application to receive the following over the 6-month intervention:
  * personalized plans for aerobic-based PA
  * personalized resistance exercise sessions
  * engagement strategies.
  Interventions: Behavioral: Digital Exercise Intervention
- Enhanced Usual Care (No Intervention): The enhanced usual care arm will receive their usual care in addition to a passive physical activity tracker device. No intervention materials will be delivered to these participants over the course of their enrollment in the study.

INTERVENTIONS:
Behavioral: Digital Exercise Intervention — Subjects randomized to the intervention arm will receive the same as the enhanced usual care arm but will be additionally exposed to: (1) personalized plans for aerobic-based PA, (2) personalized resistance exercise sessions, and (3) financial and non-financial engagement strategies. These intervention components will be delivered continuously using an advanced digital health informatics platform during the 6 months of the intervention. The intervention will be overseen and supplemented by the exercise physiologist, who will meet with participants on a weekly, then biweekly and finally monthly basis over 6 months.
  Arms: Digital Exercise Intervention

SUMMARY:
The goal of this randomized control trial is to learn about physical fitness and exercise habits in children aged 10-17 with the Fontan Circulation through a home-based, digital exercise intervention. The main questions it aims to answer are:

* Does a home-based, digital intervention increase physical activity (PA) in youth with the FC compared to enhanced usual care?
* Does a home-based, digital intervention increase physical fitness in youth with the FC compared to enhanced usual care?
* Do multi-level factors (medical, neurodevelopmental, sociodemographic, neighborhood) impact the effectiveness of the digital intervention?

Researchers will compare participants in the enhanced usual care arm to those in the exercise intervention arm to see if the digital intervention is effective.

All participants will wear a PA tracker for 12 months and complete testing at baseline, 6 months, and 12 months.

In addition, participants in the exercise intervention arm will complete a 6-month exercise intervention with the following components:

* aerobic exercise
* resistance exercise
* engagement strategies

DETAILED DESCRIPTION:
The Fontan Circulation is associated with poor exercise performance and reduced quality of life. Current standard of care encourages physical activity (PA) in this population, but few structured interventions exist. Participants will be randomly assigned to either enhanced usual care (PA tracker and standard encouragement) or an interactive digital intervention that includes personalized aerobic and resistance exercises with behavioral engagement strategies. This study will evaluate a home-based, digital intervention delivered through a mobile health platform to promote PA and improve fitness among youth with FC.

The study will recruit up to 200 participants aged 10-17 years with FC. After initial testing and a two-week run-in period, 120 participants with peak VO2 between 45% and 80% of predicted norms will be randomized. The intervention will last 6 months, followed by a 5.5-month monitoring phase. Outcomes will include changes in PA (measured via accelerometry), peak VO2, muscle strength, body composition, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Fontan Circulation present
* Girls ≥11 years of age or menstruating must have negative urine pregnancy test
* Neurodevelopmental capacity to complete all study procedures
* Physical capacity to complete all study procedures
* English speaking with at least one English speaking parent/guardian
* To enroll in the randomized control trial, percent predicted peak VO2 <80% of age-sex matched normal controls on the baseline exercise stress test (EST)

Exclusion Criteria:

* Inability to complete an EST at any time (i.e. limited physical or executive function)
* Uncontrolled lymphatic disorders
* Exercise induced or uncontrolled arrhythmias
* Pacemaker or internal cardiac defibrillator (ICD)
* Peak VO2 <45% age-sex predicted
* Having had or under consideration for a heart transplant
* Pregnant or lactating females
* Parents/guardians or subjects who, in the opinion of the investigator, may be non-compliant with study schedules or procedures

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
MIMS-units | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in total volume of physical activity (PA) operationalized as a Monitor Independent Movement Summary (MIMS) units, expressed as a percentile based on what is expected for their age and sex.
Absolute peak VO2 | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in absolute peak VO2, the maximum amount of oxygen the body consumes during exercise without regard to body weight (liters/minute).
Percent predicted peak VO2 | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in percent predicted peak VO2, the maximum amount of oxygen the body consumes during exercise expressed as a percentage of what is expected for their age and sex.
Leg lean mass | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in leg lean mass presented as a z-score. Leg lean mass z-score compares an individual's leg muscle mass to the average for their age and sex, with values below -2.0 indicating lower-than-expected muscle mass.

SECONDARY OUTCOMES:
MVPA | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in time spent in moderate to vigorous physical activity (MVPA), in terms of minutes per day.
Forearm strength | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in forearm strength measured via handgrip test and presented as a z-score. Z-scores are used to standardize measurements across individuals with different demographics (i.e. age, sex, body size).
Lower extremity strength | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in lower extremity strength measured via knee and ankle peak torsion and presented as a z-score.
PROMIS Pediatric Profile-25 T-score | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Profile-25. This 25-item questionnaire provides a T-score based on physical function, anxiety, depression, fatigue, peer relationships and pain. Children and parents will complete a PROMIS questionnaire. Children will answer questions about themselves and parents will answer questions in regard to their child.
PCQLI score | 0 to 12 months. Evaluated from baseline to 6 months, baseline to 12 months, and 6 to 12 months.
  Change in Pediatric Cardiac Quality of Life Instrument (PCQLI) total and sub-scale scores (i.e. Disease Impact, Psychosocial Impact).The PCQLI is a cardiac-specific health-related quality-of-life instrument. Children will answer questions about themselves and parents will answer questions in regard to their child.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Goldmuntz, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
NHLBI data sharing regulations will be followed. No data will be shared before study conclusion.